CLINICAL TRIAL: NCT03824782
Title: The Effect of Eyemasks on Neonatal Stress Following Dilated Retinal Examination, a Randomized Clinical Trial
Brief Title: The Effect of Eyemasks on Neonatal Stress Following Dilated Retinal Examination
Acronym: MASK-ROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Dr. Eugene Ng, Chief, Newborn & Developmental Paediatrics, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 307-2016
Record Dates: First submitted 2019-01-21; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Retinopathy of Prematurity; Pain; Premature Infant; Retinal Disease
Keywords: Retinopathy of Prematurity; ROP; Screening; Stress; Pain; Photophobia; Neonate; Light Sensitivity; Desaturation; Bradycardia; Apnea
MeSH Terms: conditions — Retinopathy of Prematurity; Pain; Premature Birth; Retinal Diseases; Photophobia; Bradycardia; Apnea

STUDY DESIGN:
Intervention Model Description: A dual-centre, prospective parallel group trial with balanced randomization (1:1) will be conducted.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Infants in the control arm received standard examinations to screen for retinopathy of prematurity.
- Standard of Care + Phototherapy Mask (Experimental): Infants in the treatment arm will have a standard phototherapy mask (Biliband, Natus, Pleasanton, California, USA) applied over the eyes after instillation of mydriatic drops. The masks will be removed 4 hours after the eye examination, when the pharmacologic effect of the mydriatic agents would have subsided. Infants will then receive standard examinations to screen for retinopathy of prematurity. The mask will be removed for the examination but reapplied promptly afterward.
  Interventions: Device: Phototherapy Mask

INTERVENTIONS:
Device: Phototherapy Mask — A standard phototherapy mask (Biliband, Natus, Pleasanton, California, USA) applied over the eyes after instillation of mydriatic drops. The masks will be removed 4 hours after the eye examination, when the pharmacologic effect of the mydriatic agents would have subsided.
  Arms: Standard of Care + Phototherapy Mask

SUMMARY:
Although screening exams for retinopathy of prematurity (ROP) prevent blindness they are physiologically stressful for infants. The investigators postulate that photosensitivity during mydriasis contributes to post-examination stress and that reducing light stimulation with a phototherapy mask can make infants more comfortable. The objective of this study is to determine the effect of a phototherapy mask worn during mydriasis on infant stress in the 12 hour period following ROP screening.

DETAILED DESCRIPTION:
Retinopathy of Prematurity (ROP) is a disorder of retinal vascular development of the low birthweight preterm infant that may lead to blindness if untreated. The long term visual acuity of infants with ROP detected by screening examination can be improved by peripheral retinal ablation therapy or injection of anti-VEGF agents.

The screening examination for retinopathy of prematurity involves dilation with mydriatic eye drops, insertion of a lid speculum to retract the eyelids, and depression of the sclera to visualize the retina. These exams are routinely performed in Neonatal Intensive Care Units (NICUs) to facilitate early detection of ROP and guide treatment to prevent retinal detachment and blindness. However, infants undergoing this examination have shown elevations in heart rate, blood pressure, and desaturations at the time of the examination, and in the hours following. The frequency of apneic events experienced by these infants is increased in the 24-48 hour period after an examination.

Several studies have looked at the pain response to mydriatic drops and speculum insertion as well as the systemic effects of the mydriatic drops. However, the cause of apneic events in the later post-examination period is unknown. The investigators postulate that photosensitivity related to mydriasis is distressing for infants in the period before and after the ROP exam, potentially contributing to stressful events, including apnea.

The investigators propose to test this hypothesis by conducting a dual-centre, prospective parallel group trial with balanced randomization (1:1), applying a phototherapy mask (Biliband, Natus, Pleasanton, California, USA) to cover the eyes of the infant after the instillation of mydriatic drops, leaving the mask on for 4 hours, the typical duration of mydriasis following a drop of cyclopentolate. The investigators expect that this intervention will result in a significant reduction in the number of stressful events following an examination, and may reduce the amount of distress experienced by infants. Infants requiring ROP screening will be automatically identified as part of routine hospital protocols. Participants will be recruited from the NICUs at St. Michael's Hospital and Sunnybrook Health Sciences Hospital in Toronto, Ontario, Canada.

The investigators predict that infants that have had their eyes shielded from environmental light while dilated are less likely to experience distressful events in the 12 hour period following ROP screening. If this study shows decreased rates of distress using this therapy, it would be a very simple addition to current practice and be of benefit for premature infants undergoing an uncomfortable exam.

ELIGIBILITY:
Inclusion Criteria:

* Infant with birthweight of ≤1500 g or less or a gestational age of ≤ 32 weeks with no prior ROP screening. Examinations will be performed starting at either 4 weeks chronological age or 31 weeks post menstrual age, whichever is later.

Exclusion Criteria:

* Pre-existing corneal abrasion/ulcers, ocular malformations that prevent dilation, and known neurological abnormalities that could affect response to pain.
* Anticipation of transfer to another institution.
* Prior ROP screening

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Number of all stressful events | 12 hours after examination
  Count of all desaturations, bradycardic events, and apneic events, adjusted for baseline rate of stressful events 12 hours prior to examination.
  Infants are under continuous vital sign monitoring and these events are flagged using the following parameters:
  Desaturation = Pulse oxymetry <88% Bradycardia = Heart rate <100bpm Apneic episode = Cessation of respiratory effort >20 seconds, or less if accompanied by bradycardia, cyanosis or pallor

SECONDARY OUTCOMES:
Number of desaturations | 12 hours
  Count of events 12 hours after examination, adjusted for baseline rate of events 12 hours prior to examination.
  Desaturation = Pulse oxymetry <88%.
Number of bradycardic events | 12 hours
  Count of events 12 hours after examination, adjusted for baseline rate of events 12 hours prior to examination.
  Bradycardia = HR < 100bpm
Number of apneic events | 12 hours
  Count of events 12 hours after examination, adjusted for baseline rate of events 12 hours prior to examination.
Heart Rate | 4 hours
  Heart Rate (bpm) recorded every hour after the ROP exam
Respiratory Rate | 4 hours
  Respiratory Rate (RPM) recorded every hour after the ROP exam
Oxygen saturation | 4 hours
  Oxygen saturation (Oximetry %) recorded every hour after the ROP exam

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Szigiato AA, Speckert M, Zielonka J, Hollamby K, Altomare F, Ng E, Nisenbaum R, Sgro M. Effect of Eye Masks on Neonatal Stress Following Dilated Retinal Examination: The MASK-ROP Randomized Clinical Trial. JAMA Ophthalmol. 2019 Nov 1;137(11):1265-1272. doi: 10.1001/jamaophthalmol.2019.3379. PMID 31486844

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT03824782/Prot_SAP_000.pdf